CLINICAL TRIAL: NCT04452383
Title: The Effect Of Adding Ketamine to Propofol For Drug-induced Sleep Endoscopy in Adult Patients With Obstructive Sleep Apnea A Randomized Controlled Study
Brief Title: f Adding Ketamine to Propofol For Drug-induced Sleep Endoscopy in Adult Patients With Obstructive Sleep Apnea
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Heba Mohamed EL -Asser,MD, principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Sedation in DISE
Record Dates: First submitted 2020-06-21; First posted 2020-06-30 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Ketamine; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A computer-generated randomization table divided patients into 2 equal groups randomly allocated patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol (P) (Active Comparator): patients will receive only propofol intravenous for sedation
  Interventions: Drug: propofol
- propofol ketamine (pk) (Active Comparator): patients will receive ketamine in addition to propofol intravenous for sedation
  Interventions: Drug: Ketamine + propofol

INTERVENTIONS:
Drug: Ketamine + propofol — effect of adding ketamine to propofol for patients undergoing DISE surgery
  Other Names: ketamine
  Arms: propofol ketamine (pk)
Drug: propofol — effect of IV propofol alone for patients undergoing DISE surgery
  Other Names: diprivan
  Arms: propofol (P)

SUMMARY:
The investigator compared the sedative effects of propofol alone and ketamine added to propofol in drug induced sleep endoscopy

DETAILED DESCRIPTION:
Propofol and ketamineare commonly used intravenous anesthetic drug used for procedural sedation.

The investigator compared the effect of propofol and propofol ketamine in patients undergoing drug induced sleep endoscopy.

ELIGIBILITY:
Inclusion Criteria

* Age > 18 years old.
* American society of anesthesiologists (ASA) physical status I or II. I / II

Exclusion Criteria:

* patient refusal
* American society of anesthesiologists (ASA) physical status > III
* known or suspected allergy to the studied drugs or its components, allergy to eggs or soy beans
* morbid obesity
* patients with moderate to severe chronic obstructive pulmonary disease or uncontrolled asthma, congestive e heart failure ,seizures ,or cerebrovascular disease
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with successful completion of the procedure (with diagnosis of site and degree of obstruction) | the duration of the procedure under sedation is usually about 20 minutes to complete the procedure
  Number of patients with successful completion of the procedure (with diagnosis of site and degree of obstruction)

SECONDARY OUTCOMES:
time until suﬃcient sedation to start endoscopy | It is about 5-10 minutes from start of studied drug till patient is ready to start endoscopy
  time to start endoscopy is deﬁned as the duration between start of the studied drugs until MOAA/S Modified observer assessment scale of alertness sedaion score 1 was obtained.
The total propofol and ketamine dose(mg)/patient needed/patient was calculated | the procedure
  The total propofol and ketamine(mg) /patient dose needed/patient was calculated
any airway intervention and occurrence of laryngospasm after start of the DISE procedure until its completion with diagnosis of site and degree of obstruction | the procedure
  Once the DISE began, the airway interventions were important as outcomes, because these interrupted the clinical study of the DISE. Furthermore, laryngospasm was deﬁned by the requirement for positive pressure ventilation of >20 cmH2O or administration of succinylcholine or propofol or any .
Adverse events (hypotension, bradycardia, arrhythmia, laryngospasm, cough, gag reﬂex, apnea or aspiration) were recorded during the procedure | the procedure
  Bradycardia was diagnosed if heart rate dropped below 60beats/min and atropine 0.01mg/kg was given if HR decreased below 50beats/min. Hypotension was diagnosed if mean arterial blood pressure (MAP) decreased by more than 30% from baseline or below 60mmHg
Time till Recovery | an average of 5 minutes between stop of drugs until Modified observer's assessment of alertness sedation MOAA/S became 4
  Time between stop of the study drugs until Modified observer's assessment of alertness sedation MOAA/S score of 4 was calculated and patient is shifted to recovery room( MOAA/S score btween 0-6 where 1 patient is ready for endoscopic airway evaluation and 1 patient is ready for discharge to recovery room ) Time till (MOAA/S) score 4 was calculated .
patients and surgeon satisfaction | about 30 minutes after complete recovery both patients' and surgeon satisfaction were recorded using a 7-point Likert-like verbal rating scales for patients and surgeon satisfaction where 7 is extremely satisfied and 1 is extremely dissatisfied
  Both patients' and surgeon satisfaction were recorded using a 7-point Likert-like verbal rating scales for patients and surgeon satisfaction where 7 is extremely satisfied and 1 is extremely dissatisfied
Time to Aldrete's recovery scores became 10 (maximum) (patient is ready to discharge) was recored post procedure in the recovery room | Average 15-30 minutes post procedure to have Aldrete's recovery scores 10 (maximum) (patient is ready to discharge) in the recovery room
  Time to Aldrete's recovery scores became 10 (maximum)(patient is ready to discharge) was recorded post procedure in the recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Heba M EL-Asser, MD, Principal Investigator — Zagazig University
Locations (1):
- zagazig University, Zagazig, Sarkia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho JS, Soh S, Kim EJ, Cho HJ, Shin S, Kim HJ, Koo BN. Comparison of three sedation regimens for drug-induced sleep endoscopy. Sleep Breath. 2015 May;19(2):711-7. doi: 10.1007/s11325-015-1127-9. Epub 2015 Feb 3. PMID 25643766
- [Background] De Vito A, Agnoletti V, Berrettini S, Piraccini E, Criscuolo A, Corso R, Campanini A, Gambale G, Vicini C. Drug-induced sleep endoscopy: conventional versus target controlled infusion techniques--a randomized controlled study. Eur Arch Otorhinolaryngol. 2011 Mar;268(3):457-62. doi: 10.1007/s00405-010-1376-y. Epub 2010 Sep 2. PMID 20811901